CLINICAL TRIAL: NCT06500403
Title: Noninvasive Tools for the Diagnosis of Porto-sinusoidal Vascular Disease: a Single-center, Prospective, Cohort Study
Brief Title: Non-invasive Tools for PSVD Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-566
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Non-Cirrhotic Portal Hypertension; Porto-Sinusoidal Vascular Diseases
MeSH Terms: conditions — Idiopathic Noncirrhotic Portal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have received platinum-based chemotherapy for organ tumors
  Interventions: Diagnostic Test: liver and stiffness measurement

INTERVENTIONS:
Diagnostic Test: liver and stiffness measurement — liver and spleen stiffness measurement are non-invasive tools for evaluation of cirrhosis and portal hypertension

SUMMARY:
Patients treated with platinum-based chemotherapy drugs have the probability of developing PSVD. The diagnosis of PSVD depends on liver biopsy. In addition, the level of portal vein pressure has guiding value in the diagnosis and prognosis of PSVD. Many studies have shown that liver and spleen stiffness have high accuracy in diagnosis and prognosis. The purpose of this study is to evaluate the efficacy of the combination of liver and spleen stiffness in the diagnosis of PSVD and to search for effective biomarkers for the diagnosis of PSVD through a single-center, prospective, observational study.

DETAILED DESCRIPTION:
PSVD is a supplement to non-cirrhotic portal hypertension and is defined as a class of diseases with characteristic pathological changes based on portal vein or hepatic sinuses abnormalities without cirrhosis. Some patients treated with platinum-based chemotherapy drugs will develop PSVD, which is clinically manifested as portal hypertension related complications. The diagnosis of PSVD depends on liver biopsy. In addition, the level of portal vein pressure has guiding value in the diagnosis and prognosis of PSVD. However, liver biopsy and pressure measurement are invasive methods. Many studies have shown that liver and spleen stiffness have high accuracy in diagnosis and prognosis. The purpose of this study is to evaluate the efficacy of the combination of liver and spleen stiffness in the diagnosis of PSVD and to search for effective biomarkers for the diagnosis of PSVD through a single-center, prospective, observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Received platinum chemotherapy for organ tumors;
2. Ages 18-80;
3. sign the informed consent voluntarily.

Exclusion Criteria:

1. Liver pathology suggested cirrhosis;
2. Underwent liver transplantation;
3. Combined with hepatocellular carcinoma exceeding Milan criteria;
4. Complicated with severe heart, kidney, or lung failure;
5. Pregnant or lactating women;
6. Data is seriously missing;
7. Patients were judged not suitable for participation in this study by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had organ tumors and had received platinum chemotherapy before, the expected survival time is not less than half of year.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Searching for valid non-invasive tools for the diagnosis of PSVD | 2 years
  The sensitivity and specificity of the non-invasive models for the diagnosis of PSVD reached 85% and 60%, respectively

SECONDARY OUTCOMES:
Patients developed portal-hypertension-related complications | 3 years
  clinically significant ascites, esophagogastric variceal hemorrhage, hepatic encephalopathy, etc.
Patients died | 3 years
  All-cause death
Patients underwent liver transplantation | 3 years
  Patients underwent liver transplantation during follow up
Patients reached the final follow-up time | 3 years
  Patients had accepted 3-year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang hospital, Southern Medical Uiversity, Guangzhou, Guangdong, China